CLINICAL TRIAL: NCT02919241
Title: An Application of Treatment Regarding a Diagnostic Interview and One-session Cognitive Behavioural Therapy - Effectiveness in Treatment of Dental Fear
Brief Title: Diagnostic Interview and One-session Cognitive Therapy in Treatment of Dental Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKuopio 001/2016
Record Dates: First submitted 2016-09-23; First posted 2016-09-29 (Estimated); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Dental Fear
Keywords: dental anxiety; cognitive therapy
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diagnostic interview (Experimental): Intervention for this group include diagnostic interview. Oral health Impact Profile (OHIP 14) and Spielberg State and Trait Anxiety (STAI-1) questionnaires and behaviour analyses are used in diagnostic interview.
  Interventions: Behavioral: Diagnostic interview
- Combined interview and treatment (Experimental): Intervention for this group include both the diagnostic interview and one session treatment.
  Interventions: Behavioral: Diagnostic interview; Behavioral: Combined interview and treatment.

INTERVENTIONS:
Behavioral: Diagnostic interview — A profound interview to declare causes for negative thoughts, assumptions and beliefs towards dental care. Participants come from public and Private dental care.
Behavioral: Combined interview and treatment. — Intervention for this group include both the diagnostic interview to declare causes for negative thoughts, assumptions and beliefs towards dental care and one session treatment. Participants come from the Institute of Dentistry.
  Arms: Combined interview and treatment

SUMMARY:
Clinical trial of an application of cognitive behavioural one-session therapy method with patients who have severe or average dental fear/anxiety measured by Modified Dental Anxiety Scale (MDAS). The intervention consists of two different parts: a diagnostic interview and one-session treatment of dental care. The method is based on One-Session Therapy manual (Öst & Skaret, 2013). 30 minimum 18 years old adults takes part to the study. They comes from three different places,primary care clinic, community dental care and dentist´s teaching clinic.

DETAILED DESCRIPTION:
Purpose is to compare diagnostic interview (n=20) to diagnostic interview and one-session treatment of dental care (n=10). Partners come from three different places, 10 from each: public and private dental care and dental school. Participants from dental school take part to one-session treatment. All participants have normal dental care before final interview. Hypotheses is that dental fear/anxiety will decrease one category (5 points) when measured by Modified dental anxiety scale (MDAS) before the intervention and after normal dental care. Visual Analogue Scale is used to measure the strength of unpleasant feeling before and after intervention in both groups.

ELIGIBILITY:
Inclusion Criteria:

* MDAS 13 or over, dental care in normal circumstances doesn´t work, motivation to treat dental fear, minimum 18 year

Exclusion Criteria:

* Mental disorder, dementia, pregnancy, acute state of somatic illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-08; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in dental fear | 6 months
  Change in fear is measured by a questionnaire called Modified Dental Anxiety Scale (MDAS). Change in fear is indicated by change in mean value of the MDAS between baseline and follow-up measurement

SECONDARY OUTCOMES:
Compliance to care | 6 months
  Compliance to care is indicated if treatment defined before the baseline interview can be wholly executed. If patient interrupt treatment or cannot be executed at all after baseline interview, then compliance is not fulfilled.

CONTACTS AND LOCATIONS:
Overall Officials: Liisa Suominen, Professor, Study Director — University of easthern Finland, Kuopio
Locations (1):
- University of Eastern Finland, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No
It has been planned to use same data later in a follow-up study

REFERENCES:
- [Derived] Kurki P, Korhonen M, Honkalampi K, Suominen AL. Patients' multifaceted views of dental fear in a diagnostic interview. Acta Odontol Scand. 2021 Apr;79(3):194-204. doi: 10.1080/00016357.2020.1817545. Epub 2020 Sep 12. PMID 32924725